CLINICAL TRIAL: NCT02181049
Title: Cardiac and Vascular Late Sequelae in Long-term Survivors of Childhood Cancer (CVSS): a Multidisciplinary Clinical, Epidemiological and Genetic Approach
Brief Title: Cardiac and Vascular Late Sequelae in Long-term Survivors of Childhood Cancer (CVSS)
Acronym: CVSS
Status: Active, not recruiting | Type: Observational
Sponsor: CVSS study (Other)
Collaborators: Univ. Prof. Dr. med. Joerg Faber, Center for Pediatrics, Hematology, Oncology and Hemostaseology (Unknown); Univ. Prof. Dr. med. Philipp S. Wild, MSc, Preventive Cardiology and Preventive Medicine, Center for Cardiology, Clinical Epidemiology, CTH (Unknown); Dr. oec. troph. Hiltrud Merzenich, Insitute for Medical Biometry, Epidemiology and Informatics (IMBEI) (Unknown)
Responsible Party: Sponsor-Investigator, CVSS study, interdisciplinary cooperation, Johannes Gutenberg University Mainz
Organization: Johannes Gutenberg University Mainz (Other)
Other Study IDs: CVSS-study
Record Dates: First submitted 2014-06-27; First posted 2014-07-03 (Estimated); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Childhood and Adolescence Cancer (Survivors and Deceased)
Keywords: Childhood cancer survivors; Cardiac; Vascular; Cardiovascular; Late-sequelae
MeSH Terms: conditions — Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — blood, serum, plasma, DNA, RNA, urine, tear fluid
Oversight: Data Monitoring Committee: No

SUMMARY:
Due to remarkable advances in childhood cancer therapy the 10-year survival rate increased to over 80% and late sequelae come to the fore. Childhood cancer survivors (CCS) suffer from significant excess in mortality risk associated with treatment-related complications at least for 25 years after the initial cancer diagnosis. In particular, the prevalence of cardiovascular disease seems to be elevated compared to the general population. The CVSS study is a multi-disciplinary cooperation project between the Institute for Medical Biostatistics, Epidemiology and Informatics (IMBEI) and the German Childhood Cancer Registry (GCCR), the Preventive Cardiology and Preventive Medicine and the Pediatric Hematology and Oncology all at the University Medical Center of the Johannes Gutenberg University Mainz. The central element is a thorough clinical cardiovascular examination of all patients, which permits detecting subclinical disease. Therapy data will be extracted retrospectively from various sources. The study intends to describe the current situation of a cohort of approximately 1000 CCS in Germany aged 24 to 49 years with respect to cardiovascular health. The role of risk factors (treatment related and classic cardiovascular risk factors), as well as related predisposing genetic factors is investigated. The results will contribute to recommendations to improve follow-up care.

ELIGIBILITY:
Inclusion Criteria:

1. Survivors of oncological disease according to ICCC-3 aged <15 years at diagnosis, diagnosed 1980-1990 while resident in Germany
2. Declaration of consent for storage of personal data at GCCR

Exclusion Criteria:

1. Patient has refused contact with GCCR
2. Current address not available
3. Second malignant neoplasm
4. Diagnosis Morbus Hodgkin
5. Diagnosis WILMS tumor in 1990
6. Former treating center recommends exclusion
7. Insufficient knowledge of German language
8. Inability to travel to the study center and participate in the examinations

Ages: 24 Years to 49 Years | Sex: All
Age Groups: Adult
Study Population: Survivors of a oncological disease according to ICCC-3 aged <15 years at diagnosis, diagnosed 1980-1990 while resident in Germany
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Heart failure | up to 35 years after exposure to childhood cancer therapy
Hypertension | up to 35 years after exposure to childhood cancer therapy

SECONDARY OUTCOMES:
Myocardial infarction | up to 35 years after exposure to childhood cancer therapy
Late-occurring stroke | up to 35 years after exposure to childhood cancer therapy
  "late" is defined as 5 years or more after diagnosis of cancer
Carotid artery disease | up to 35 years after exposure to childhood cancer therapy

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Faber, Univ.-Prof. Dr. med., Principal Investigator — Center for Pediatrics, Pediatric Hematology, Oncology and Hemostaseology, University Medical Center of the Johannes Gutenberg University Mainz; Philipp S Wild, Univ.-Prof. Dr. med. MSc, Principal Investigator — Preventive Cardiology and Preventive Medicine, Center for Cardiology, Clinical Epidemiology, Center for Thrombosis and Hemostasis (CTH), University Medical Center of the Johannes Gutenberg University Mainz; Hiltrud Merzenich, Dr. oec. troph., Principal Investigator — Institute for Medical Biostatistics, Epidemiology and Informatics (IMBEI), University Medical Center of the Johannes Gutenberg University Mainz
Locations (1):
- University Medical Center of the Johannes Gutenberg University Mainz, Mainz, Rhineland-Palatinate, Germany

REFERENCES:
- [Derived] Arnold N, Merzenich H, Wingerter A, Schulz A, Schneider A, Prochaska JH, Gobel S, Neu MA, Henninger N, Panova-Noeva M, Eckerle S, Spix C, Schmidtmann I, Lackner KJ, Beutel ME, Pfeiffer N, Munzel T, Faber J, Wild PS. Promotion of Arterial Stiffness by Childhood Cancer and Its Characteristics in Adult Long-Term Survivors. J Am Heart Assoc. 2021 Feb;10(5):e015609. doi: 10.1161/JAHA.119.015609. Epub 2021 Feb 24. PMID 33624513